CLINICAL TRIAL: NCT03348527
Title: A Single Blind, Two-Stage Dose Finding Study to Evaluate the Safety, Tolerability and Efficacy of a Single Liproca® Depot Injection Into the Prostate in Patients With Localized Prostate Cancer, Assigned to Active Surveillance Who Are at High Risk for Disease Progression (Followed by an Open Label Extension With a Repeat Injection (Optional)).
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of a Liproca® Depot Injection in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lidds AB (Industry)
Collaborators: CMX Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LPC-004
Record Dates: First submitted 2017-11-01; First posted 2017-11-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Stage I: 20 Subjects will be enrolled into one of two groups, each receiving a single dose of Liproca®Depot. The target treatment dose will be 35% (Cohort 1) or 45% (Cohort 2) of the prostate volume (mL).
  Stage II: 40 subjects will be randomized to receive either 16 mL (Cohort 3) or 20mL (Cohort 4) of Liproca®Depot.
Who Masked: Participant
Masking Description: Participant is blinded to whether they are receiving a treatment dose of 35% or 45% of total prostate volume in stage I or 16mL or 20mL in stage II.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage I: Dose = 35% of prostate volume (Experimental): Subject will be randomized into a group receiving one dose of 2-hydroxyflutamide depot (Liproca® Depot) equal to 35 % of their prostate volume.
  Interventions: Drug: 2-Hydroxyflutamide Depot
- Stage I: Dose = 45% of prostate volume (Experimental): Subject will be randomized into a group receiving one dose of 2-hydroxyflutamide depot (Liproca® Depot) equal to 45 % of their prostate volume.
  Interventions: Drug: 2-Hydroxyflutamide Depot
- Stage II: Dose = 16mL (Experimental): Subject will be randomized into a group receiving one dose of 2-hydroxyflutamide depot (Liproca® Depot) equal to 16mL
  Interventions: Drug: 2-Hydroxyflutamide Depot
- Stage II: Dose = 20mL (Experimental): Subject will be randomized into a group receiving one dose of 2-hydroxyflutamide depot (Liproca® Depot) equal to 20mL
  Interventions: Drug: 2-Hydroxyflutamide Depot

INTERVENTIONS:
Drug: 2-Hydroxyflutamide Depot — Liproca® Depot is a depot formulation containing a bioresorbable, controlled-release,formulation of the nonsteroidal antiandrogen 2-hydroxyflutamide
  Other Names: Liproca® Depot Injection

SUMMARY:
A Single Blind, Two-Stage Dose Finding Study to Evaluate the Safety, Tolerability and Efficacy of a Single Liproca® Depot Injection into the Prostate in Patients with Localized Prostate Cancer,Assigned to Active Surveillance who are at High Risk for Disease Progression (followed by an Open Label Extension with a Repeat Injection (Optional))

DETAILED DESCRIPTION:
Patients assigned to Active Surveillance and who have fulfilled all inclusion criteria will receive a prophylactic antibiotic and a local anaesthetic (according to the Investigator's Standard of Care) prior to administration of Liproca® Depot.

60 subjects will be enrolled.

The Single Dose Study will be conducted in two stages:

In Stage I, 20 subjects will be randomized into two groups to receive one dose of Liproca® Depot equal to 35% (Cohort 1) or 45 % (Cohort 2) of their prostate volume (mL) (N=10:10). Two weeks after all subjects have received their initial dose, the Data Safety Monitoring Board (DSMB) will review the subjects' safety and tolerability data over the first 14 days after receiving treatment.

In Stage II, 40 subjects will be randomized to receive either 16mL (Cohort 3) or 20mL (Cohort 4) of Liproca® Depot.

All subjects in Stage I and Stage II will be followed for 24 weeks.

Subjects who complete the Single Dose Study and who experience no safety or tolerability issues, as determined by the Investigator, may be offered an option to participate in the Open Label Extension Study (OLE). Subjects enrolled in the OLE will be observed for PSA recurrence every 8 weeks. If PSA recurrence is confirmed (defined as a PSA level exceeding at least 100 % of Baseline value) subjects will receive a second treatment of Liproca® Depot. The dose will be injected into the tumour focus/foci and in close proximity to the tumour, based on a prostate biopsy (and MRI, if applicable), using a TRUS for guidance.

Stage I subjects who received 35% volume of Liproca® Depot will receive 16 mL and subjects who received 45% volume of Liproca® Depot will receive 20 mL. Stage II subjects will receive the same dose of Liproca® Depot that was administered in the first treatment.

Subjects in the OLE receiving a second injection will be followed up for an additional 24 weeks for safety, tolerability and efficacy. After this period, subjects may undergo MRI imaging and a prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study specific procedures being performed
* 18 - 80 years of age, inclusive
* Assigned to Active Surveillance
* Histologically confirmed, localized prostate cancer within 24 months of Screening
* Gleason score 3+3 or 3+4 with one or more of the following characteristics:

PSA > 6.0 μg/L (ng/mL) and PSA density > 0.15; PSA > 10.0 μg/L and < 20 μg/L (ng/mL); Any systematic core > 50% involvement; Any PI-RADS score 4 or 5 on MRI; Any Gleason grade 4, Men of African descent

* Patient has a negative bone scan within the last 12 months
* Patient is able to have an MRI
* Prostate volume ≤ 80 mL (measured by MRI within 12 months of Screening or has been scheduled for an MRI prior to Screening)
* eGFR ≥ 30 mL/min, using the Cockcroft - Gault Equation: = [{(140 - age in years) x (weight in kg)} x 1.23] / serum Creatinine in micromol/l
* AST, ALT and ALP ≤ 1.5 times upper limit of normal
* Patient must be willing to comply with all study procedures
* Patients must agree to the use of medically acceptable methods of contraception, including non-hormonal intrauterine device (IUD) or double barrier method (condom with foam or vaginal spermicidal suppository, diaphragm with spermicide) for the duration of the study (24 weeks), unless the patient and/or their partner has been surgically sterilized

Exclusion Criteria:

* PSA > 20 μg/L (ng/mL)
* Previous or ongoing hormonal therapy for prostate cancer
* Positive urine culture before treatment with prophylactic antibiotics
* Ongoing or previous therapy with finasteride or dutasteride in the last 3 months
* Ongoing or previous invasive therapy for benign prostate hyperplasia (BPH) (e.g. TURP,TUMT, HIFU, etc.)
* Use of pacemaker or other implanted electronic devices
* Metal implant in the pelvis (e.g. hip replacement) that may affect the MRI of the prostate
* Allergy to Liproca® Depot and its ingredients
* Severe micturition symptoms (I-PSS >15 or residual urine volume > 150 mL) confirmed by repeat measurement or Qmax< 12 mL/s
* Ongoing therapy with the anticoagulant Acetyl Salicylic Acid (ASA) (more than 100mg/day) as preventive anti-thrombotic therapy should be withdrawn temporarily before treatment with Liproca® Depot, as determined by the Investigator. Other anticoagulants should be withdrawn in cooperation with the treating physician
* Use of any previous focal prostate cancer treatment, such as transurethral resection, cryotherapy, high intensity frequency ultrasound (HIFU) and/or photodynamic therapy
* Concomitant systemic treatment with corticosteroids or immune modulating agents
* Known immunosuppressive disease (e.g. HIV, Type II Diabetes). Patients with well controlled Type II Diabetes may be included, as determined by Investigator
* Simultaneous participation in any other study involving an investigational product or device,or having participated in a prostate cancer study within the last 12 months prior to starting treatment with Liproca® Depot
* Infection in WHO Risk Group 2, 3 or 4

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Highest Tolerable Dose of Liproca Depot | 24 weeks
  To define the highest tolerable dose of Liproca Depot for transrectal injection into the prostate.

SECONDARY OUTCOMES:
Liproca Depot Effect on Prostate Specific Antigen Levels | 24 weeks
  To determine the absolute level and % decrease of PSA level at Week 8, 16, 20 and 24, and PSA nadir.
Liproca Depot Effect on Prostate Volume | 20 weeks
  To determine the effect on prostate volume at Week 20 after treatment with one of four doses of Liproca Depot based on an MRI evaluation. Measured by %decrease versus Baseline and as absolute values.
Evaluation of Lesions | 20 weeks
  MRI evaluation of Lesions based on PI-RADS (Prostate Imaging Reporting and Data System) score 20 weeks after treatment with one of four doses of Liproca Depot.
Quality of Life (QoL) Questionnaire Score | 24 weeks
  Assessment of QoL Questionnaire scores at Baseline, Week 8,16,20 and 24 after treatment with one of four doses of Liproca Depot.
Micturition Status using the International Prostate Symptom Score (I-PSS) | 24 weeks
  Micturition status will be assessed using the I-PSS Questionnaire at Week 8, 20 and 24 after treatment with one of four doses of Liproca Depot.
Frequency of Adverse Events | 24 weeks
  All adverse events related to Liproca Depot or its administration, incidence of AEs, withdrawals due to AEs and all Serious Adverse Events (SAEs) will be assessed. All adverse events will be reported and followed until resolved or until, in the Investigator's opinion, the condition has become stable and is unlikely to change further.
Change in Testosterone Levels | 24 weeks
  Testosterone levels (nmol/L) will be assessed at Baseline, Week 8 and 24 after treatment with one of four doses of Liproca Depot.
Systematic Exposure of 2-hydroxyflutamide | 24 weeks
  To examine the systematic exposure of 2-hydroxyflutamide at Baseline, Hour 2, Day 2,4,7 and 14, week 8 and end of study for all subjects in Phase I and a subset of 12 subjects in Stage II.
Pharmacokinetics of 2-hydroxyflutamide | 24 weeks
  To examine the pharmacokinetics of 2-hydroxyflutamide at Baseline, Hour 2, Day 2,4,7 and 14, week 8 and end of study for all subjects in Phase I and a subset of 12 subjects in Stage II.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Casey, MD, Study Director — CMX Research
Locations (10):
- Canada (6):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Jonathan Giddens Medicine Professional Corporation, Brampton, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences, Kaunas
  - National Cancer Institute - Oncourology Department, Vilnius